CLINICAL TRIAL: NCT06928168
Title: Effect of Sleep Extension in Prevention to Sleep Deprivation on Running Endurance Performance
Brief Title: Effect of Sleep Extension in Prevention to Sleep Deprivation
Acronym: SLEEPERF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Jean Monnet University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 24CH296; 2024-A02857-40 (Other: ANSM)
Record Dates: First submitted 2025-03-28; First posted 2025-04-15 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Healthy
Keywords: Sleep deprivation; Sleep extension; Endurance running; Fatigue
MeSH Terms: conditions — Sleep Deprivation; Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- REP (reproducibility). (Experimental): This group will perform an incremental running test, driven to exhaustion, after a night of total sleep deprivation twice, at least two weeks apart.
  Interventions: Other: Reproductibility
- PT (total sleep deprivation). (Experimental): This group will perform an incremental running test, conducted until exhaustion, in:
  * a control condition (usual sleep)
  * a one-night condition of partial sleep deprivation
  * a one-night partial sleep deprivation condition with 5 nights of prior extension. The order of conditions will be randomized.
  Interventions: Other: Total sleep deprivation
- PP (partial sleep deprivation) (Experimental): This group will perform an incremental running test, run to exhaustion, in :
  * a control condition (usual sleep),
  * a one-night total sleep deprivation condition
  * a one-night total sleep deprivation condition with 5 nights of extension beforehand. The order of conditions will be randomized.
  Interventions: Other: partial sleep deprivation

INTERVENTIONS:
Other: Total sleep deprivation — This group will perform an incremental running test, conducted until exhaustion, in: - a control condition (usual sleep) - a one-night condition of partial sleep deprivation - a one-night partial sleep deprivation condition with 5 nights of prior extension. The order of conditions will be randomized.
  Arms: PT (total sleep deprivation).
Other: partial sleep deprivation — This group will perform an incremental running test, conducted until exhaustion, in: - a control condition (usual sleep) - a one-night condition of partial sleep deprivation - a one-night partial sleep deprivation condition with 5 nights of prior extension. The order of conditions will be randomized.
  Arms: PP (partial sleep deprivation)
Other: Reproductibility — This group will perform an incremental running test, driven to exhaustion, after a night of total sleep deprivation twice, at least two weeks apart.
  Arms: REP (reproducibility).

SUMMARY:
The approach of a competition can be associated to a decrease in sleep duration and quality which can negatively impact athlete's performance and health (injury risk, fall, accident). Ultra-endurance competitions even involve partial and/or total sleep deprivation over one or several nights. Studied investigating this question suggest that endurance performance under sleep deprivation is altered, mainly because of an effect on the rate of perceived exertion (RPE), which regulates effort intensity. One of the methods used by athletes to limit the impact of sleep deprivation in competition is to implement sleep extension in the days prior to a competition. However, few studies have investigated the impact of sleep deprivation et its reproducibility on performance and fatigue during a prolonged running exercise, as well as the efficiency of prior sleep extension. The importance of such a preventive measure might also depend on individual resistance to sleep deprivation, which is variable between persons and could have genetic determinants. This aspect remains under-studied, particularly regarding the impact of sleep deprivation on physical performance. Therefore, this study aims at investigating the effects of sleep deprivation and prior sleep extension on prolonged duration performance.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer who signed the written consent form.
* Man or woman.
* Aged 18-50.
* Physically active and running at least one session of more than one hour per week.
* Haven't participated in any competition in the month before the first visit.
* Not participating in any competition during the study.
* Usual sleep time between 6h-8h per night.

Exclusion Criteria:

* - Any chronic pathology.
* Working night shift.
* Having sleep disorders: score > 5 at Pittsburg Sleep Quality Index.
* Excessive sleepiness: score >10 at Epworth Sleepiness scale.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 69 (Estimated)
Dates: Start 2025-06-12 (Actual); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Performance over a standardized incremental running test | Day 7
  Sporting performance, measured by the duration of exercise in a time-limited incremental effort test in running to exhaustion, i.e. the inability to maintain the imposed pace.

SECONDARY OUTCOMES:
Reproducibility of sleep deprivation effects. | Day 7
  Repeatability of sleep deprivation effects will be assessed within the REP group by comparing performance on the time limit test (in minutes) after each sleep deprivation.
Resistance to sleep deprivation and genetic polymorphism | DAy 1
  The influence of genetic polymorphism will be evaluated via the effects of sleep deprivation according to the genetic polymorphism of the ADORA2A, TNFα and COMT genes
Fatigue (objective and subjective, ) | DAy 7
  Neuromuscular fatigue will be assessed by the loss of isometric knee extensor muscle strength measured before and just after the time limit test. To characterize the origin of neuromuscular fatigue, electrically evoked forces from peripheral nerve stimulation and electrical muscle activity (EMG) will be measured to quantify central and peripheral fatigue.
Fatigue (sleepiness) | DAy 7
  Sleepiness will be assessed using the Epworth Sleepiness Scale, and perceived exertion will be rated on a Borg scale from 6 to 20 during submaximal exercise prior to the time limit test, and regularly during the test.
Fatigue (perception of effort) | DAy 7
  Perceived fatigue will be rated on a 0-10 scale before and after the time limit test.
Motor function (running biomechanics ) | Day 7
  Motor function will be assessed during 40 minutes of submaximal exercise at an intensity corresponding to the first ventilatory threshold (SV1) preceding the time limit test. Running biomechanics will be investigated by measuring ground reaction forces (in Newtons) using force platforms integrated into an instrumented treadmill.
Motor function (energy cost) | Day 7
  Motor function will be assessed during 40 minutes of submaximal exercise at an intensity corresponding to the first ventilatory threshold (SV1) preceding the time limit test. The energy cost of running (Cr, in J/kg/m) will be quantified by measuring gas exchanges over a 5-minute period.
Cognitive function (vigilance) | Day 7
  Cognitive function will be assessed before, during and after exercise using Psychomotor Vigilance Task (PVT)
Cognitive function (attention) | Day 7
  Cognitive function will be assessed before, during and after exercise using concentration test (sustained attention task).
Cognitive function (inhibition) | Day 7
  Cognitive function will be assessed before, during and after exercise using a battery of tests including inhibition test (Go-no Go task)

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric ROCHE, PhD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- FEASSON Léonard, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No
this study involves a small number of subjects and is taking place only in ST-ETIENNE